CLINICAL TRIAL: NCT07156383
Title: Effects of CBT-I on Hypothalamic-Pituitary-Adrenal (HPA)-Axis Functioning in Participants With Chronic Insomnia
Brief Title: Restorative Effects of Sleep on Everyday Health and Wellbeing: A Treatment Study
Acronym: RESET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Responsible Party: Principal Investigator, Ivan Vargas, Assistant Professor, University of Notre Dame
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-01-9063
Record Dates: First submitted 2025-08-20; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Insomnia
Keywords: Sleep Initiation and Maintenance Disorders; Insomnia Disorder; Sleep Disorders; Cortisol; Sleep Deprivation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Sleep Deprivation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A within, between subjects design will be used with a four week run-in period (to establish a baseline) prior to the intervention phase (randomly assigned to one of two active interventions that are administered in parallel).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-Week CBT-I (Experimental): Participants in this arm will receive 4 weeks of CBT-I.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- 10-Week CBT-I (Experimental): Participants in this arm will receive 10 weeks of CBT-I.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia (CBT-I) is the first line treatment for Insomnia. Participants will receive weekly CBT-I during which they will receive the tools to improve their sleep.

SUMMARY:
The purpose of this study is to evaluate the mechanisms through which Cognitive Behavioral Therapy for Insomnia (CBT-I) leads to improvements in sleep and sleep-related daytime outcomes, specifically as it relates to cortisol and the hypothalamic-pituitary-adrenal (HPA) axis, the body's primary stress response system. The primary research aims are: 1) To determine whether changes in cortisol functioning are related to improvements in sleep consolidation (4-week CBT-I), sleep duration (10-week CBT-I) or both, AND 2) to examine whether these improvements are more pronounced among individuals with insomnia and short sleep duration (compared to insomnia with 'normal' sleep duration).This study will recruit individuals with chronic insomnia: half with reported short sleep duration (less than 6 hours of sleep on an average night) and half with reported non-short sleep duration (6 or more hours per night). Participants will complete an in-lab assessment on four different occasions. During the first visit, they will confirm eligibility, complete an online survey, complete an in-lab stress task (with saliva samples), and provide a hair sample to measure cortisol (a hormone). They will then be sent home with a home sleep test as a final eligibility check (to rule out sleep disorders other than insomnia), an actigraphy watch to measure their sleep, and collection tubes to provide saliva samples to measure cortisol. We will then track the participants' sleep using online daily diaries and actigraphy for four week. Following the 4-week baseline period, participants will come in for a second in-lab visit (same procedures as the first visit) and then be randomized to receive either four or ten weeks of Cognitive Behavioral Therapy for Insomnia (CBT-I). CBT-I is a empirically supported behavioral treatment for insomnia and the first-line treatment for chronic insomnia. Sleep patterns and insomnia symptoms will continue to be monitored via diaries during the intervention phase. The third visit will take place once the participant has completed the intervention and the fourth visit will occur three months following the third visit (3 months post-treatment). The 3rd and 4th visits will again replicate the same procedures conducted during the initial lab visit.

ELIGIBILITY:
Inclusion Criteria:

* At least 18-years-old
* Speaks English
* Meets DSM-5 criteria for Insomnia Disorder, determined through initial screener than verified during brief clinical interview (at intake)

Exclusion Criteria:

* Sleep disorders other than Insomnia
* Endocrine disorders
* Extreme sleep schedule (i.e. shift workers)
* Currently taking sleep medication
* Currently taking medication for endocrine dysfunction
* Currently taking medication that interferes with sleep or cortisol levels
* Excessive alcohol/substance use or AUD/SUD
* Serious mental illness
* Chronic medical conditions (which may be exacerbated by sleep restriction)
* Pregnant or nursing women
* Women in the peri-menopausal stage due to irregular menses and fluctuations in sex hormones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Symptoms | From enrollment through study completion - up to 7 months depending on assigned treatment group. Measured at Baseline, Pre-treatment, Post-Treatment, and Follow-Up (end of study).
  Total score on the Insomnia Severity Index (ISI), which ranges from 0-28. Higher scores indicate greater insomnia severity, while lower scores indicate less insomnia severity.
Sleep Continuity Disturbance | From enrollment through study completion - up to 7 months depending on assigned treatment group. Measured at Baseline, Pre-treatment, Post-Treatment, and Follow-Up (end of study).
  Mean sleep latency, wake after sleep onset, and early morning awakenings (in minutes assessed via daily sleep diaries).
Total Sleep Time | From enrollment through study completion - up to 7 months depending on assigned treatment group. Measured at Baseline, Pre-treatment, Post-Treatment, and Follow-Up (end of study).
  Mean sleep duration (in minutes) assessed via daily sleep diaries
HPA-Axis Functioning | From enrollment through study completion - up to 7 months depending on assigned treatment group. Measured at Baseline, Pre-treatment, Post-Treatment, and Follow-Up (end of study).
  Salivary cortisol assessed in three ways: hair (chronic stressor exposure), at-home saliva (basal cortisol), and saliva in response to an in-lab stressor (stress reactivity).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Notre Dame, Notre Dame, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available upon completion of the study and publication of the study results. These data will be made available online through a dedicated study site.
Supporting Information: Study Protocol, Analytic Code
Time Frame: De-identified IPD will be made available indefinitely upon publication of the primary study results.